CLINICAL TRIAL: NCT07197554
Title: A Phase 1/1B Study of ST-01156, a Small Molecule RBM39 Degrader, in Patients With Advanced Solid Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SEED Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST-01156-101
Record Dates: First submitted 2025-08-28; First posted 2025-09-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumors; Ewing Sarcoma; Hepatocellular Carcinoma (HCC); Biliary Tract Cancer (BTC)
Keywords: cancer; solid tumors; RBM39; RBM39 degrader; metastatic solid malignancies; Ewing sarcoma; Hepatocellular carcinoma; HCC; Biliary tract carcinoma; endometrial carcinoma; Adolescents
MeSH Terms: conditions — Sarcoma, Ewing; Carcinoma, Hepatocellular; Biliary Tract Neoplasms; Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): ST-01156, administered orally once daily for 5 consecutive days followed by 2 days without study drug administration every 7 days
  Interventions: Drug: ST-01156

INTERVENTIONS:
Drug: ST-01156 — ST-01156 is an orally administered degrader of RBM39, a protein frequently upregulated in cancer

SUMMARY:
A Phase 1/1B Study of ST-01156 in Patients with Advanced Solid Malignancies

DETAILED DESCRIPTION:
This Phase 1/1b study is evaluating the safety, tolerability, and preliminary anticancer activity of ST-01156 in participants with advanced solid malignancies. The study will be conducted in 2 parts. Part 1 (Dose Escalation) will assess the safety, tolerability, pharmacokinetics (PK) and preliminary anticancer activity of SD-01156 in participants with advanced solid malignancies, many of whom have a biological rationale to be targeted with an inhibitor of RBM39. Part 1 will also seek to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of ST-01156.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years on the day of signing the consent form, except for adolescents with Ewing Sarcoma or other malignancies for which there is a biological rationale to support participation, in which case the participant is ≥ 16 years old.
* Has a metastatic or locally advanced and unresectable solid tumor.
* Has at least 1 measurable lesion or evaluable disease per RECIST v1.1.
* Has an ECOG performance status ≤ 2 at screening.
* Has adequate organ function as defined in the protocol.

Exclusion Criteria:

* Has received prior radiotherapy within 2 weeks of treatment.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate, provided they are radiologically stable
* Has received treatment with any local or systemic anticancer therapy or investigational anticancer agent within 14 days or 5 half-lives, whichever is shorter.
* Had major surgery within 28 days before study therapy administration
* Has toxicities from previous anticancer therapies that have not resolved to baseline levels, with the exception of alopecia and peripheral neuropathy.
* Has previously received a RBM39 inhibitor/degrader.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 171 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: Dose Escalation | First 28 days of treatment
  To characterize the safety, tolerability, and adverse event (AE) profile of escalating doses of ST-01156 administered for 5 consecutive days followed by 2 days without study drug administration every 7 days, with a cycle defined as 28 days (4 weeks).
Part 1: Dose Escalation | Duration of treatment period
  To identify the maximum tolerated dose (MTD) or maximum administered dose (MAD), and to recommend a dose for subsequent studies (recommended Phase 2 dose [ RP2D]) of ST-01156 on a daily oral schedule for 5 consecutive days out of every 7 days with a cycle defined as 28 days (4 weeks).

SECONDARY OUTCOMES:
Part 1: Dose Escalation | First 28 days of treatment
  To characterize the pharmacokinetics (PK) of ST-01156 administered on a daily oral schedule for 5 consecutive days every 7 days with cycle defined as 28 days (4 weeks). PK parameters will include area under the concentration-time curve (AUC), maximum observed concentration (Cmax), and time to observe maximum observed concentration (Tmax).
Part 1: Dose Escalation | Baseline and every 6 weeks thereafter until disease progression
  To detect preliminary evidence of antitumor activity in select advanced cancers where strong preclinical evidence of the anticancer activity of RBM39 degradation is strongest including:
  * Adults or adolescents with ES following disease progression or intolerance to therapeutics of reasonable likelihood of conferring clinical benefit.
  * aHCC following disease progression or intolerance to appropriate standard therapy for advanced disease.
  * KRASm solid malignancy of any type - locally advanced or unresectable solid malignancy following disease progression or intolerance to therapeutics or reasonable likelihood of conferring clinical benefit.
  * BTC, endometrial carcinoma, solid malignancies with pathogenic somatic or germline mutations in BCRA1/2 or HRR genes (BRCA1/2, PALB2, RAD51C, RAD51D, ATM, BARD1, BLM, BRIP 1, CDK12,FANCA, FANCC, FANCD2, FANCE, FANCF, FANCM, MRE11A, NBN (NBS1), RAD50, RAD51B and others as confirmed by a Clinical Laboratory Improvement Amendments [CLIA]-certified m

OTHER OUTCOMES:
Part 1: Dose Escalation | Days 1, 2, 3, 4, 5, 8, 15, and 16 of the first two 28-day cycles of treatment, and days 1 of subsequent cycles, until permanent discontinuation of study treatment.
  To evaluate the relationship between RBM39 degradation in peripheral blood mononuclear cells (PBMC) [and potentially other cells or tissues], to various safety and efficacy endpoints.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - The City of Hope National Medical Center, Duarte, California
  - Hoag Memorial Hospital, Newport Beach, California
  - Mass General Brigham Cancer Institute, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No